CLINICAL TRIAL: NCT00361660
Title: The Impact of Functional Task Practice Dosing on Motor Control in Hemiplegia From Chronic Stroke
Brief Title: The Effect of Different Schedules of Functional Task Practice for Improving Hand and Arm Function After Stroke
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: project was only internally funded and would complete for subjects with 2 newer externally funded projects
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Richards, Lorie - Principal Investigator, Department of Veterans Affairs
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 407-2005A
Record Dates: First submitted 2006-08-07; First posted 2006-08-08 (Estimated); Last update posted 2015-06-26 (Estimated); Status verified 2015-06

CONDITIONS: Cerebrovascular Accident; Hemiplegia
Keywords: Motor skills; Occupational Therapy; Physical Therapy Techniques; Rehabilitation; Upper Extremity; Stroke
MeSH Terms: conditions — Stroke; Hemiplegia | interventions — Constraint Induced Movement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Therapy is provided every other day 3 days per week (Monday, Wednesday, Friday).
  Interventions: Behavioral: functional task practice - distributed
- 2 (Active Comparator): The same therapy is provided daily Monday through Friday
  Interventions: Behavioral: functional task practice - condensed

INTERVENTIONS:
Behavioral: functional task practice - distributed — This functional task practice is modeled after Constraint-Induced Movement Therapy in which participants wear a mitt on the non-paretic arm for up to 90% of waking hours and then attend therapy for 3 hours a session Monday, Wednesday, and Friday in which they practice various functional tasks, such as tracing a stencil, placing toothbrushes in toothbrush holders, etc.
  Other Names: constraint-Induced Movement Therapy
  Arms: 1
Behavioral: functional task practice - condensed — This functional task practice is modeled after Constraint-Induced Movement Therapy in which participants wear a mitt on the non-paretic arm for up to 90% of waking hours and then attend therapy for 3 hours a session Monday through Friday in which they practice various functional tasks, such as tracing a stencil, placing toothbrushes in toothbrush holders, etc.
  Other Names: Constraint-Induced Movement Therapy
  Arms: 2

SUMMARY:
The first purpose of this study is to determine how often people should practice motor skills to best improve the ability to use the affected arm and hand after stroke. The second purpose is to determine whether it is better to practice a lot of repetitions of a few tasks or a few repetitions of many tasks during motor rehabilitation for the arm and hand after stroke.

DETAILED DESCRIPTION:
Intense skill practice with the affected arm after stroke has the potential to improve upper extremity (UE) function resulting from neuroplastic changes in the motor cortex. However, the necessary and sufficient parameters of this therapy in humans have not been fully investigated. Delineation of the most efficacious and efficient therapy for promoting UE recovery post-stroke is necessary before effective clinical implementation of this therapy. In this study, using parallel group design methodology, we will test the effect of 2 practice parameter (i.e. spacing of practice and number of repetitions per task practiced per session) modifications on UE function following skill practice.

Forty subjects will complete multiple baseline testing and then be randomized, using random number table, to one of 4 groups: condensed functional task practice modeled after Constraint-Induced Movement Therapy (6 hours of practice/day, 5 days/week, 2 weeks), condensed functional task practice with a restricted number of tasks practiced, distributed, distributed functional task practice (Monday, Wednesday, Friday, 6 hours/session, 10 sessions), distributed functional task practice with a restricted number of tasks practiced. During therapy sessions, subjects will practice performing common activities with their paretic upper extremity. They will wear a mitt on their non-paretic upper extremity for up to 90% of their waking hours. Post-testing sessions will follow within one week of completing therapy with an additional follow-up testing session 3 months later.

ELIGIBILITY:
Inclusion Criteria:

* hemiparesis due to unilateral stroke at least 3 months prior
* 18-90 years of age
* able to extend the paretic wrist 200 and at least 1 finger 100
* able to follow 2-step commands
* score < 3 on the Motor Activity Log Amount of Use scale

Exclusion Criteria:

* have no medical or orthopedic condition that would significantly limit ability to participate in the intervention or benefit from the therapy
* have no history of other major neurologic or psychiatric condition or injury, and have no active drug or alcohol abuse.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-08; Primary Completion 2007-08 (Actual); Study Completion 2007-12 (Estimated)

PRIMARY OUTCOMES:
Upper extremity subscale of the Fugl-Meyer Motor Assessment | immediately after therapy ends

SECONDARY OUTCOMES:
Wolf Motor Function Test | Immediately after therapy ends

CONTACTS AND LOCATIONS:
Overall Officials: Lorie G Richards, PhD, Principal Investigator — North Florida/South Georgia Veterans Health System